CLINICAL TRIAL: NCT01543854
Title: A Multicenter, Double Blind, Randomized, Parallel Group, Placebo-controlled Study to Evaluate the Hemodynamic Responses to Intravenous RLX030 Infusion in Subjects With Acute Heart Failure
Brief Title: Hemodynamic Responses to RLX030 Infusion in Subjects With Acute Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRLX030A2201; 2011-000833-35 (EudraCT Number)
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Acute Heart Failure
Keywords: Heart failure; RLX030; Hemodynamics; Cardiovascular Diseases
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases | interventions — serelaxin protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- RLX030 (Experimental): RLX030 as intravenous infusion for 20 hours
  Interventions: Drug: RLX030
- Placebo (Placebo Comparator): Matching placebo as intravenous infusion for 20 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RLX030 — Intravenous infusion of RLX030 over 20 hrs
  Other Names: serelaxin*; *International Nonproprietary Name
  Arms: RLX030
Drug: Placebo — Intravenous infusion of placebo over 20 hours
  Arms: Placebo

SUMMARY:
This study will assess the hemodynamic effect of RLX030 infusion in subjects with acute heart failure. In addition safety and effects on renal function and biomarkers will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized or requiring admission to hospital for management of acute heart failure within the previous 48 hours.
* Pulmonary wedge pressure above or equal to18 mmHg determined by right heart catheterization

Exclusion Criteria:

* Systolic blood pressure below 115 mmHg
* Significant valvular diseases or arrythmias
* Acute coronary syndrome in previous 45 days
* Treatment with mechanical support (intra-aortic balloon pump, endotracheal intubation, mechanical ventilation, or any ventricular assist device)
* Impaired renal or hepatic function

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Peak change from baseline of PCWP (pulmonary capillary wedge pressure) | baseline, after 8 and 20 hrs treatment
  Measurements will be made using a Swan-Ganz indwelling catheter
Peak change from baseline of CI (cardiac index) | baseline, after 8 and 20 hrs treatment
  Measurements will be made using a Swan-Ganz indwelling catheter

SECONDARY OUTCOMES:
Change over time of PCWP (pulmonary capillary wedge pressure) | During 20 hours of infusion and up to 4 hours after stop of infusion
  Measurements will be made using a Swan-Ganz indwelling catheter
Change over time of systemic vascular resistance (SVR) | During 20 hours of infusion and up to 4 hours after stop of infusion
  Measurements will be made using a Swan-Ganz indwelling catheter
Change over time of pulmonary vascular resistance (PVR) | During 20 hours of infusion and up to 4 hours after stop of infusion
  Measurements will be made using a Swan-Ganz indwelling catheter
Change over time of pulmonary arterial pressure (PAP) | During 20 hours of infusion and up to 4 hours after stop of infusion
  Hemodynamic measurements were made using a Swan-Ganz catheter when patients were in a supine position
Change over time of pulmonary and peripheral oxygen saturation | During 20 hours of infusion and up to 4 hours after stop of infusion
  Hemodynamic measurements were made using a Swan-Ganz catheter when patients were in a supine position
Pharmacokinetics of RLX030: area under the serum concentration-time curve from time zero to infinity (AUCinf) | During 20 hours of infusion and 24 hours after stop of infusion
  Blood will be collected from an in dwelling catheter.
Pharmacokinetics of RLX030: area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) | During 20 hours of infusion and 24 hours after stop of infusion
  Blood will be collected from an in dwelling catheter.
Pharmacokinetics of RLX030: serum concentration over 20 hours of infusion (C20h) | During 20 hours of infusion and 24 hours after stop of infusion
  Blood will be collected from an in dwelling catheter.
Pharmacokinetics of RLX030: terminal elimination half-life (T1/2) | During 20 hours of infusion and 24 hours after stop of infusion
  Blood will be collected from an in dwelling catheter.
Pharmacokinetics of RLX030: mean residence time (MRT) | During 20 hours of infusion and 24 hours after stop of infusion
  Blood will be collected from an in dwelling catheter.
Pharmacokinetics of RLX030: volume of distribution at steady state following intravenous administration | During 20 hours of infusion and 24 hours after stop of infusion
  Blood will be collected from an in dwelling catheter.
Change over time on calculated creatinine clearance | During 20 hours of infusion and 4 hours after stop of infusion
  Urine samples will be collected for analyses.
Change over time in Diuresis | During 20 hours of infusion and 4 hours after stop of infusion
  Urine samples will be collected for analyses.
Central aortic systolic pressure-time curve | During 20 hours of infusion and 24 hours after stop of infusion
  A cuff will be used for a brachial blood pressure measurement and a wrist sensor for arterial pulse waveforms
Radial augmentation index-time curve | During 20 hours of infusion and 24 hours after stop of infusion
  A cuff will be used for a brachial blood pressure measurement and a wrist sensor for arterial pulse waveforms
Number of patients with adverse events, serious adverse events and death | During 20 hours of infusion and 24 hours after stop of infusion
  Adverse events will be assessed by signs/symptoms, clinical laboratory and electrocardiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- Argentina (2):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
- Germany (6):
  - Novartis Investigative Site, Bad Nauheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Halle
- Novartis Investigative Site, Brescia, BS, Italy
- Novartis Investigative Site, Groningen, Netherlands
- Poland (2):
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Russia (5):
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, S.-Petersburg
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Tomsk

REFERENCES:
- [Derived] Ponikowski P, Mitrovic V, Ruda M, Fernandez A, Voors AA, Vishnevsky A, Cotter G, Milo O, Laessing U, Zhang Y, Dahlke M, Zymlinski R, Metra M. A randomized, double-blind, placebo-controlled, multicentre study to assess haemodynamic effects of serelaxin in patients with acute heart failure. Eur Heart J. 2014 Feb;35(7):431-41. doi: 10.1093/eurheartj/eht459. Epub 2013 Nov 18. PMID 24255129